CLINICAL TRIAL: NCT01276548
Title: A Trial to Evaluate Efficacy and Safety of the Combination Therapy of Genexol®-PM Plus Carboplatin® Compared to Genexol® Plus Carboplatin® as a Firstline Treatment in Subjects With Ovarian Cancer
Acronym: GPMOC202
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samyang Biopharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GPMOC202
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Genexol®-PM plus Carboplatin (Experimental)
  Interventions: Drug: Genexol®-PM 260mg/m2 plus Carboplatin 5 AUC
- Genexol® plus Carboplatin (Active Comparator)
  Interventions: Drug: Genexol® 175mg/m2 plus Carboplatin 5 AUC

INTERVENTIONS:
Drug: Genexol®-PM 260mg/m2 plus Carboplatin 5 AUC
  Arms: Genexol®-PM plus Carboplatin
Drug: Genexol® 175mg/m2 plus Carboplatin 5 AUC
  Arms: Genexol® plus Carboplatin

SUMMARY:
The purpose of this study is to Evaluate Efficacy and Safety of the Combination Therapy of Genexol®-PM Plus Carboplatin® Compared to Genexol® Plus Carboplatin® as a Firstline Treatment in Subjects With Ovarian Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who aged 18 years or older
2. Subjects whose written informed consent was obtained complying with the local regulatory requirements prior to their participation in the trial
3. Subjects who have histologically or cytologically confirmed unresectable or metastatic epithelial cancer of the exocrine pancreas. High-quality contrast-enhanced CT scanning is required to evaluate resectability. Measurable disease is not required.

Exclusion Criteria:

1. Subjects who have received prior radiation therapy (XRT) for pancreatic cancer unless progression was documented after XRT and 6 weeks have elapsed between completion of XRT and start of trial medication.
2. Subjects who have had systemic treatment such as chemotherapy or immunotherapy, for pancreatic cancer. However, prior use of chemotherapy, e.g. 5-FU or capecitabine, for radiation sensitization is allowed. If gemcitabine was given in the adjuvant setting, only subjects relapsed with cancer after 6 months of completing the last dose of gemcitabine can participate in the trial.
3. Subjects who have had a major surgery within 2 weeks prior to the screening/baseline visit

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2009-10; Primary Completion 2012-05 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of Genexol®-PM plus Carboplatin versus Genexol® plus Carboplatin in subjects with ovarian cancer based on Composite Response Rate | up to 6 cycles
  Proportion of subjects with CA125 and RECIST composite response rate was evaluated and compared between the groups. CA125 was evaluated among subjects without a measurable disease, while RECIST was evaluated among subjects with a measurable disease; discordance between the response rates by RECIST and CA125 were deemed as nonresponse.

SECONDARY OUTCOMES:
Overall Survival | up to 3 years
  The period from the date of first administration to the date of the patient's death
Progression Free Survival | up to 3 years
  The period from the date of first administration to the date of objective tumor progression by CA125 and RECIST or death
Time to Progression | up to 3 years
  The period from the date of first administration to the date of tumor progression by CA125 and RECIST or objective tumor progression, excluding progression-free death

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, Pungnap-2 Dong, South Korea